CLINICAL TRIAL: NCT00260182
Title: Genetics of Recurrent Early Onset Major Depression
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas F. Levinson, Principle Investigator, Stanford University
Other Study IDs: R01MH061686-02 (NIH); R01MH061686-02 (NIH); R01MH059542 (NIH); R01MH059552 (NIH); R01MH075131 (NIH); R01MH059541 (NIH); R01MH060912 (NIH); DNBBS 7G-GRR
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: Depressive Disorder; Family; Genetics
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples with DNA

SUMMARY:
This study will identify specific genes that may cause a predisposition to depression in some families.

DETAILED DESCRIPTION:
Depression is a serious medical illness that is often difficult to diagnose and treat. Studies on patterns of depression within families suggest that inherited genes may cause a predisposition to the disorder. People with early onset depression often have more relatives with depression than people whose depression does not begin until later in life. It is likely that several interacting genes cause this tendency towards the disorder, rather than one specific gene. This study will serve to identify particular genes that may cause a susceptibility to depression in order to better understand the brain mechanisms involved with severe depression. In turn, this may aid in the development of new treatments for depression.

Participation in this observational study will entail one interview and one blood test. Participants will be interviewed, either in person or by telephone, about their personal and family psychiatric history. The blood sample will be collected at a time and location that is convenient for the participant. Participants may also be asked to invite other family members to participate in the study.

For information on a related study please follow this link:

http://clinicaltrials.gov/show/NCT00005914

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent major depression
* Has a parent or sibling with a history of recurrent major depression
* Depression began before the age of 31

Exclusion Criteria:

* Bipolar I (manic-depressive) disorder
* Schizophrenia

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include participants with a family history of depression.
Sampling Method: Non-Probability Sample
Enrollment: 2302 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Major depressive disorder diagnosis | One patient interview session (typically 2 hours), and blood draw (10-20 minutes)
  The study will correlate genome-wide SNP genotypes with case vs. control status, defined by presence or absence of major depressive disorder.
  Participants will attend an interview regarding personal and family history of psychiatric disorders, and give a blood specimen. Genotypes from blood samples will be studied for association with presence of major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas F. Levinson, MD, Principal Investigator — Stanford University; Myrna M. Weissman, PhD, Principal Investigator — Columbia University/New York State Psychiatric Institute; J. Raymond DePaulo, MD, Principal Investigator — Johns Hopkins University; William A. Scheftner, MD, Principal Investigator — Rush University Medical Center; William Coryell, MD, Principal Investigator — University of Iowa; William Lawson, MD, Principal Investigator — Howard University
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - Howard University, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University/New York State Psychiatric Institute, New York, New York

REFERENCES:
- See also: Click here for the Stanford University study web page — http://depressiongenetics.stanford.edu